CLINICAL TRIAL: NCT04930640
Title: A 8 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of SGF200 on Immune Enhancement
Brief Title: The Efficacy and Safety of SGF200 on Immune Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BL-PI-SGF200
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Immunity
Keywords: SGF200

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGF200 group (Experimental): 1 times a day, 1 capsule for 1 time, before breakfast meal[350 mg/day (Bacillus amyloliquefaciens spore 1x10^9 CFU/day, GF101 200 U/day)]
  Interventions: Dietary Supplement: SGF200 group
- placebo group (Placebo Comparator): 1 times a day, 1 capsule for 1 time, before breakfast meal[350 mg/day (Bacillus amyloliquefaciens spore 0 CFU/day, GF101 0 U/day)]
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SGF200 group — 1 times a day, 1 capsule for 1 time, before breakfast meal, for 8 week
  Arms: SGF200 group
Dietary Supplement: Placebo — Placebo for 8 week
  Arms: placebo group

SUMMARY:
This study was conducted to investigate the efficacy and safety of SGF200 on immune enhancement.

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled human trial. 100 subjects were randomly divided into SGF200 group or placebo group. The investigators measured Natural Killer cell activity, Cytokines(IL-2, IL-12, IFN-γ, TNF-α), questionnaire scores of upper airway infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 50 years
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* If screening shows that the white blood cell(WBC) is less than 3000/㎕ or more than 8000/㎕
* Those who received influenza vaccination within 3 months before first intake for test product
* Those who have a body mass index(BMI) of less than 18.5 kg / m^2 or greater than 35 kg / m^2 at the screening
* Those who have a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry, musculoskeletal system, inflammatory and hematologic
* Those who take a medication or health function food that affects your promotion of immunity within 1 month prior to the screening
* Those who have received antipsychotic medication within 3 months before screening
* Those who alcoholic or drug abuse suspected
* Those who participated in other clinical trials within 3 months before screening
* Laboratory test by show the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Changes of Natural Killer cell activity | 8 weeks
  Natural Killer cell activity was measured in study baseline and 8 week. A ratio of effector cell and target cell was 2.5:1, 5:1, 10:1
  (Experimental - Effector Spontaneous - Target Spontaneous) / (Target Maximum - Target Spontaneous) × 100

SECONDARY OUTCOMES:
Changes of Cytokines | 8 weeks
  For blood Cytokines analysis, collect 3 ml of blood in one SST tube for 5 ml, leave at room temperature for 30 minutes for clotting, after then centrifuge at 3000 rpm (or 2000 xg) for 10 minutes.
  Inspection item were IL-2, IL-12, IFN-γ, TNF-α.
Changes of Wisconsin Upper Respiratory Symptom Survey-21 | 8 weeks
  Wisconsin Upper Respiratory Symptom Survey-21 consists of seven steps, including individual symptoms, functional quality of life, and overall improvement. Find the sum of the symptom questions and give them the total score. Seek, sum up the questions of life, and get the total quality of life. The sum of the total score of symptoms and the total score of quality of life is also obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea